CLINICAL TRIAL: NCT06893718
Title: Effects of Treadmill Training With and Without Compression Stockings on Toe Walking and Balance in Children With Autism.
Brief Title: Treadmill Training With and Without Compression Stockings on Toe Walking and Balance in Children With Autism.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/qutbia abaq
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: "Autism, Toe Walking, Treadmill, Compression Stockings.
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A intervention: Compressions Stocking Group (Experimental): * Duration:
  * Stockings for 1 hour before and during treadmill walking.
  * Treadmill for 10 minutes.
  * Frequency: 5 sessions/ week for 6 weeks.
  Interventions: Other: Compressions Stocking Group; Other: Treadmill Training Group
- Group B intervention: Treadmill Training Group (Active Comparator): Duration: Treadmill for 10 minutes.
  • Frequency: 5 sessions/ week for 6 weeks.
  Interventions: Other: Compressions Stocking Group; Other: Treadmill Training Group

INTERVENTIONS:
Other: Compressions Stocking Group — * Incline: Initially 5% incline and after 4 weeks an incline of 10% will be observed
  * Speed: Constant speed of 3.4 mph.
  * Warm up: Calf stretch 10 reps/ 2 sets.
Other: Treadmill Training Group — * Incline: Initially 5% incline and after 4 weeks an incline of 10% will be observed
  * Speed: Constant speed of 3.4 mph.
  * Warm up: Calf stretch 10 reps/ 2 sets.

SUMMARY:
Autism Spectrum Disorder (ASD) affects around 1.7% of US children, with co-occurring conditions like ADHD, anxiety, and epilepsy complicating daily functioning. Early intervention strategies, such as sensory-based therapies and physical exercises like treadmill training, are used to improve motor skills and overall functioning in children with ASD. A randomized controlled trial is being conducted to evaluate the impact of treadmill interventions on children with toe-walking behaviors. Participants will be assigned to either Group A or Group B, with treadmill sessions with or without compression stockings. The study aims to investigate the potential benefits of treadmill therapy as part of a multidisciplinary approach to treating ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a complex neurodevelopmental condition characterized by difficulties in social communication, repetitive behaviors, and sensory sensitivities, typically appearing early in life. The disorder's prevalence varies globally, with recent estimates in the US showing approximately 1.7% of children affected. Diagnosis relies on comprehensive evaluations using standardized tools, such as the Autism Diagnostic Observation Schedule, to assess behavioral patterns and developmental history. Individuals with ASD often experience cooccurring conditions like ADHD, anxiety, and epilepsy, which can further impact daily functioning. Motor abnormalities, including toe-walking, are observed in some cases and may indicate underlying neurological issues or developmental delays. Early intervention, including sensory-based therapies and physical exercises like treadmill training, aims to improve motor skills and overall functioning in children with ASD, highlighting the importance of multidisciplinary support for optimal developmental outcomes.

The study will be a Randomized Controlled Trial (RCT) designed to investigate the impact of treadmill interventions on children with autism spectrum disorder (ASD) who exhibit toe-walking behaviors. Legal guardians will receive comprehensive information about the research objectives, methods, and potential benefits, and informed consent will be obtained prior to participation. Initial assessments will thoroughly evaluate each participant's baseline strength, frequency of toe walking, and balance using standardized tools like the 50-foot walk test for toe walking and the Pediatric Balance Scale for balance assessment. Participants meeting specific inclusion criteria: children diagnosed with ASD, displaying toe walking more than 30% of the time, and compliant with the treatment protocol and Exclusion Criteria: Associated orthopedic conditions, underlying genetic disorders, global developmental delay, patient's parents'/guardians' refusal to provide informed consent will be assigned to either Group A or Group B by Non- Probability Convenient Sampling technique. Group A will undergo treadmill sessions while wearing compression stockings for one hour before and during a 10-minute treadmill walk, with incline adjustments from 10% to 12% over six weeks. Group B will undergo identical treadmill sessions without compression stockings. The study will be conducted in a controlled environment at a single autism center, ensuring consistent conditions for both groups. IBM SPSS Statistics version 27 will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children with ASD who toe walk.
* Gait disorder more than 30% of the time.
* Compliance with our treatment protocol.
* Children whose guardians agreed on the study

Exclusion Criteria:

* Associated orthopedic conditions.
* Underlying genetic disorders.
* Global developmental delay.
* Patient's parents'/guardians' refusal to provide informed consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Pediatric Balance Scale | baseline, 3rd week, 6th week.
  The 14-item Pediatric Balance Scale (PBS) is a tool used to assess children's functional balance. The PBS was created by altering the Berg Balance Scale (BBS) to be used with children with cerebral palsy (CP) who have trouble responding to external stimuli and maintaining their posture. For kids with mild to severe motor impairments, the PBS has been further refined as a balancing assessment tool.
Toe Walking | baseline, 3rd week, 6th week.
  Trials frequently use the 50-Foot Timed Walk (50FTW) as a gait assessment tool. Initially, exercise-based research was the main application of the 50FWT. Around 15.24 meters (50 feet) away, the participants walk a straight line at their typical walking pace. A fat, colored tape was used to measure a distance of 15.24 meters to chart the course.

CONTACTS AND LOCATIONS:
Overall Officials: Qutbia Abaq Javed Cheema, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Asif Javed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehghani M, Jafarnezhadgero AA, Darvishani MA, Aali S, Granacher U. Effects of an 8-week multimodal exercise program on ground reaction forces and plantar pressure during walking in boys with autism spectrum disorder. Trials. 2023 Mar 8;24(1):170. doi: 10.1186/s13063-023-07158-7. PMID 36890589
- [Background] Grandits JB, Kent HW, Sanborn SM, Pilcher JJ. The effect of compression on repetitive behaviors and task participation in children with autism spectrum disorder. Front Psychol. 2023 Dec 13;14:1292439. doi: 10.3389/fpsyg.2023.1292439. eCollection 2023. PMID 38162972